CLINICAL TRIAL: NCT04529057
Title: Evaluation of the Effect of Different Rapid Maxillary Expansion Appliances on Airway by Acoustic Rhinometry: A Randomized Clinical Trial
Brief Title: Evaluation of the Effect of Different Rapid Maxillary Expansion Appliances on Airway by Acoustic Rhinometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Gökçenur Gökçe, Assistant professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDR-SABE-0024
Record Dates: First submitted 2020-08-21; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Posterior Crossbite, Upper Airway
Keywords: Rapid maxillary expansion, posterior crossbite, acoustic rhinometry

STUDY DESIGN:
Intervention Model Description: 3-arm parallel trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tooth-borne (Hyrax) expander (Experimental)
  Interventions: Procedure: Rapid Maxillary Expansion Treatment
- Tooth tissue-borne (KBME) expander (Experimental)
  Interventions: Procedure: Rapid Maxillary Expansion Treatment
- Bone-borne (MIDME) expander (Experimental)
  Interventions: Procedure: Rapid Maxillary Expansion Treatment

INTERVENTIONS:
Procedure: Rapid Maxillary Expansion Treatment — The patients were treated with KBME, Hyrax and MIDME maxillary expansion appliances, respectively. All expansion appliances containing a Hyrax expansion screw positioned parallel to the second premolars and were used to correct the posterior crossbite. In the MIDME group, two mini-screws with a diameter of 1.6 mm and a length of 10 mm are located on the right and left sides between the roots of the 2nd premolar and 1st molar teeth with 60-70° angle. KBME and Hyrax expansion appliances were cemented with glass ionomer cement and MIDME was cemented with using the light-cured composite. Same protocol was applied to all patients during RME treatment. Expansion screws in all groups were activated by two turns a day.

SUMMARY:
Rapid maxillary expansion (RME) is an orthodontic treatment based on the principle of opening the midpalatal suture with the effect of orthopedic forces. The aim of this randomized clinical study was to evaluate and compare the effects of tooth-borne, tooth-tissue borne, and bone-borne rapid maxillary expanders on nasal airway by using AR. The null hypothesis was that there is no difference for the effect on nasal airway between the appliances.

DETAILED DESCRIPTION:
Introduction: The aim of this 3-arm parallel trial was to compare the effects of tooth-borne (Hyrax), tooth tissue-borne (KBME) and bone-borne (MIDME) rapid maxillary expansion (RME) appliances on nasal airway with acoustic rhinometry (AR).

Methods: Fourty-six 12- to 14-years-old patients with narrow maxilla were randomly allocated into 3 study groups according to the type of RME appliance: tooth-borne, tooth tissue-borne and bone-borne. Participants were recruited from the Department of Orthodontics, Faculty of Dentistry, Izmir Katip Celebi University, Turkey. During the RME treatment, the same protocol was applied to all patients and the expansion screws were activated twice a day (0.4 mm/day). Computer-generated randomization was used with group allocation concealed using opaque, sealed envelopes. The outcome assessor was blinded; however, it was not feasible to blind either operator or patients. The primary outcome of this study was the correction of posterior crossbite. Secondary outcomes included AR assessment of nasal airway dimensions as nasal volume, the minimal cross-sectional area (MCA) 1 and 2. AR measurements were obtained before treatment (T0), after active expansion (T1), and at 3 months-follow-up (T2). One-way analysis of variance (ANOVA) and a Bonferroni test was used for inter-group comparison and two-way ANOVA was used for intra-group evalaution.

ELIGIBILITY:
Inclusion Criteria:

1. no previous tonsillar, nasal or adenoid surgery and orthodontic treatment,
2. Bilateral crossbite and need for RME,
3. maxillary and mandibular permanent teeth fully erupted,
4. willingness to participate in the study

Exclusion Criteria:

1. the presence of adenotonsillectomy due to tonsillar hypertrophy or adenoidal hypertrophy
2. having nasal/nasopharyngeal /oropharyngeal pathologies, craniofacial syndromes, systemic disease, poor oral hygiene,
3. history of previous orthodontic treatment.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Correction of posterior crossbite | After active expansion (up to 3 weeks) (T1).
  The palatal cusps of the maxillary posterior teeth approximated the lingual cusps of the mandibular posterior teeth.

SECONDARY OUTCOMES:
Increasing nasal cavity area-1 | At baseline (T0), after active expansion (up to 3 weeks) (T1) and after 3 months retention period (T2)
  Increasing Minimum cross-sectional area1 (MCA1)
Increasing nasal cavity area-2 | At baseline (T0), after active expansion (up to 3 weeks) (T1) and after 3 months retention period (T2)
  Minimum cross-sectional area2 (MCA2)
Increasing nasal cavity volume | At baseline (T0), after active expansion (up to 3 weeks) (T1) and after 3 months retention period (T2)
  Volume (Vol)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gokce G, Gode S, Ozturk A, Kirazli T, Veli I. Evaluation of the effects of different rapid maxillary expansion appliances on airway by acoustic rhinometry: A randomized clinical trial. Int J Pediatr Otorhinolaryngol. 2022 Apr;155:111074. doi: 10.1016/j.ijporl.2022.111074. Epub 2022 Feb 15. PMID 35189449